CLINICAL TRIAL: NCT05923502
Title: (CHANT)A Prospective, Multicenter, Non-interventionistic Real-world Study of Duvelisib Capsules in the Treatment of Non-Hodgkin's Lymphoma (NHL).
Brief Title: (CHANT)Real World Study of Duvelisib in the Treatment of Non-Hodgkin's Lymphoma (NHL)
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Ruijin Hospital
Other Study IDs: CSPC-PI3K-NHL-K01
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Follicular Lymphoma; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Richter Syndrome; Marginal Zone Lymphoma; Peripheral T Cell Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: NHL; Duvelisib
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — duvelisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All enrolled patients.: All patient who signed the consent form for participation to the study.
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — This is a real-word. The treatment options are individualized according to the diagnosis and treatment experience of doctors in each center, diagnosis and treatment specifications and individual conditions of patients.
  Other Names: Copiktra

SUMMARY:
This is a multicenter, non-interventional and prospective real-world study to evaluate the efficacy and safety of Duvelisib capsules in patients with non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional and prospective real-world study to evaluate the efficacy and safety of Duvelisib administered to subjects who have been diagnosed with non-Hodgkin's lymphoma that is relapsed or refractory, including but not limited to the following subtypes : a) Follicular lymphoma(FL); b) Chronic lymphocytic leukemia/small lymphocytic lymphoma or Richter syndrome(CLL/SLL or RS); c) Marginal zone lymphoma(MZL); d) Peripheral T-cell lymphoma(PTCL); e) Diffuse large B-cell lymphoma(DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* To participate in the study voluntarily and sign the informed consent (ICF), with good compliance and cooperative visits;
* Patients must be ≥ 18 years of age (Based on the date of signing the informed Consent (ICF));
* Pathologically or Histologically confirmed NHL including but not limited to the following subtypes:

  1. Follicular lymphoma (FL);
  2. Chronic lymphocytic leukemia/small lymphocytic lymphoma or Richter syndrome (CLL/SLL or RS);
  3. Marginal zone lymphoma (MZL);
  4. Peripheral T-cell lymphoma (PTCL);
  5. Diffuse large B-cell lymphoma (DLBCL).
* Patients who have received at least one systemic chemotherapy and have relapsed at the end of the treatment or progressed during treatment;
* Must have adequate organ function defined by the following laboratory parameters:

  1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 0.5 × 10^9/L, Platelet count (PLT) ≥ 25 × 10^9/L, blood transfusion can be used before medication;
  2. Liver and kidney function: Aspartate transaminase (AST) and alanine aminotransferase (ALT)≤5.0 × ULN;
  3. Estimated creatinine clearance value ≥30 milliliters/minute (as determined by the Cockcroft-Gault method).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Patients with infections should be treated first and then considered for enrollment when the infection is under control.

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding;
* Estimated lifetime is less than 3 months;
* In the investigator's judgment, patients who require but are unable to receive prophylactic treatment for Pneumocystis or herpes simplex virus (HSV) prior to trial drug treatment;
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function;
* Prior history of drug-induced colitis or drug-induced interstitial pneumonia;
* Known hypersensitivity to Duvelisib or its excipients;
* Administration of medications or foods that are strong inhibitors or inducers of CYP3A beginning 2 weeks prior to the first dose of Duvelisib;
* According to the judgement of the researcher, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population who have been diagnosed with non-Hodgkin's lymphoma that is relapsed or refractory, including but not limited to the following subtypes : a) Follicular lymphoma(FL); b) Chronic lymphocytic leukemia/small lymphocytic lymphoma or Richter syndrome(CLL/SLL or RS); c) Marginal zone lymphoma(MZL); d) Peripheral T-cell lymphoma(PTCL); e) Diffuse large B-cell lymphoma(DLBCL).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | From the first day of medication to 30 days after the last dose]
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 6 cycles of therapy (each cycle is 28 days)]
  Defined as the best response of complete response/remission (CR) or partial response/remission (PR).
Duration of remission (DOR) | 4 year
  Time from reaching CR or PR for the first time to disease progression.
Progression-Free-Survival (PFS) | 4 year
  From date of inclusion to date of progression, relapse, or death from any cause.
Overall survival (OS) | 4 year
  From the date of inclusion to date of death, irrespective of cause.
Quality of life (QOL) | 4 year
  The quality of life scale, ranging from 0 to 100. A score of 0 represents the worst health and a score of 100 represents the best health.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, PhD, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: Undecided